CLINICAL TRIAL: NCT05322915
Title: Therapeutic Effects of Line Dancing in People With Multiple Sclerosis: an Evaluator-blinded, Randomized Controlled Study
Brief Title: Therapeutic Effects of Line Dancing in People With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Hacettepe University (Other); Fenerbahce University (Other)
Responsible Party: Principal Investigator, FATOS KIRTEKE, PhD, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hacettepe Ergotherapy
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis
Keywords: line dance; balance; anxiety; depression; quality of life; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dance group (Experimental): The dance group, each patient received a goal-oriented line dancing program.
  Interventions: Other: line dancing
- control (No Intervention): The control group did not receive any treatment program during this period.

INTERVENTIONS:
Other: line dancing — The intervention included 60-minute sessions, two days a week for four weeks for a total of eight sessions. All sessions were administered by the physiotherapist who has 26 years of experience in dance therapy. The dance was performed on a one to one basis with minimal support from the therapist. The line dancing sequence, which was specially created for this training program, was designed as a structured goal-oriented dance. Line dancing movements/steps are comprised of moving forward and backward, or sideways and turns and scuff. In addition, the fact that one foot is always in contact with the ground makes it ideal for patients with multiple sclerosis, who may have balance problems.
  Arms: dance group

SUMMARY:
The objective of this study is to analyze the effects of line dancing on balance, anxiety, depression and quality of life for people with multiple sclerosis (PwMS).

DETAILED DESCRIPTION:
Purpose: The objective of this study is to analyze the effects of line dancing on balance, anxiety, depression and quality of life for people with multiple sclerosis (PwMS).

Methods: This study was conducted prospective parallel-group design study. 31 PwMS were randomized two groups. The dance group undertook 60-minute sessions twice a week for four weeks and the control group did not do any particular training during this period. The outcome were measured using the Berg Balance Scale (BBS), Hospital Anxiety and Depression Scale (HADS), and Multiple Sclerosis Quality of Life-54 (MSQoL-54) by an evaluator blinded to the study.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-65 years,
* EDSS [22]<6,
* Mini-Mental State Examination score >24.

Exclusion Criteria:

* exacerbations within the previous three months,
* have other physical, neurological problems,
* changeable health status.
* havig a cardiovascular disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 4 weeks
  On the scale which consists of 14 questions, individuals are given points between 0 and 4 for each question. High scores indicate good balance and low scores indicate poor balance (41-56=independent, 21-40=walks with assistance, 0-20=dependent)

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | 4 weeks
  The scale consists of 14 items, 7 of which investigate symptoms of anxiety and 7 of which investigate symptoms of depression. The scale is evaluated between 0-3 points. The cut-off value for anxiety is 10/11, and the cut-off value for depression is 7/8.
Multiple Sclerosis Quality of Life-54 | 4 weeks
  It was developed specifically to assess the quality of life of PwMS. It includes 12 parts and 54 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Ekici Çağlar, Prof, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There isn't a plan to make IPD and related data dictionaries available.